CLINICAL TRIAL: NCT03251391
Title: To Assess the Safety and Feasibility of a Structured Cardiac Rehabilitation Program in Patients With Peripheral Arterial Disease After Successful Revascularization Procedures: A Pilot Study.
Brief Title: Cardiac Rehabilitation Program in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140692
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Peripheral Arterial Disease
Keywords: revascularization; blocked arteries; leg arteries; leg pain
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation Group (Experimental): Participants randomized to this group will undergo cardiac rehabilitation program.
  Interventions: Other: Cardiac Rehabilitation Program
- Control Group (Active Comparator): Participants randomized to this group will receive care for their condition, conventional therapy, that they would normally receive.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Cardiac Rehabilitation Program — Program will involve 36 sessions. These will be scheduled as 3 sessions per week. If you cannot complete 3 sessions per week the 36 sessions could be spread out over 6 months.
  Each session will last between 30-60 minutes. Sessions will involve aerobic activity, diet/nutritional counseling, and smoking cessation information.
  Arms: Cardiac Rehabilitation Group
Other: Conventional Therapy — Participants will be asked to complete tests and questionnaires that would normally be done for their condition.
  Arms: Control Group

SUMMARY:
The main purpose of this study is to see if it is safe and feasible to use cardiac rehabilitation (CR) in patients with peripheral arterial disease (PAD) after successful revascularization. This study will also test if CR improves quality of life and health outcomes in PAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAD post-revascularization (stent, angioplasty, or bypass).
* Patients must have the ability to ambulate safely without assistance and should not have plans for undergoing further staged revascularization procedures.

Exclusion Criteria:

* Below or above the knee amputation.
* Underlying cardiopulmonary or other co-morbidity that would be an exclusion under currently approved standard CR protocols at the University of Kansas Medical Center (KUMC).
* Unfavorable short term prognosis and limited life expectancy (<2 years)
* Awaiting a planned staged revascularization in same or other leg (patients will be eligible once no further procedures are planned).
* Prior history of having dropped out of CR without completing.
* Unwilling to consent for all aspects of CR or study participation.
* Unable to come for CR (this will exclude patients who live far away or have no means to travel to the CR facility).
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-05-11 (Actual); Study Completion 2019-05-11 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk test | Change from Baseline to Up to 6 Months
  Results will be measured in meters.

SECONDARY OUTCOMES:
Short Form Health Survey 36 (SF-36) | Change from Baseline to Up to 6 Months
  Change in quality of life measured using the SF-36. The survey has 36 questions and measure eight health dimensions. The scores range from 0-100. A higher score represents less disability. A lower score represents more disability.
Short Form Health Survey 36 (SF-36) | Change from Baseline to Week 18
  Change in quality of life measured using the SF-36. The survey has 36 questions and measure eight health dimensions. The scores range from 0-100. A higher score represents less disability. A lower score represents more disability.
Vascular Quality of Life Questionnaire-6 (VascuQol6) | Change from Baseline to Up to 6 Months
  The six-item Vascular Quality of Life (VascuQol-6) is a valid, practical, and responsive instrument for the assessment of health-related QOL in patients with PAD. The main advantage is the compact format that offers a possibility for routine use in busy clinical settings.
  Range of scores and what they represent: Each question is scored 1-4. The total score is achieved by summarizing the score on each question, resulting in a score between 6 and 24. Higher value indicates better health status.
Vascular Quality of Life Questionnaire-6 (VascuQol6) | Change from Baseline to Week 18
  The six-item Vascular Quality of Life (VascuQol-6) is a valid, practical, and responsive instrument for the assessment of health-related QOL in patients with PAD. The main advantage is the compact format that offers a possibility for routine use in busy clinical settings.
  Range of scores and what they represent: Each question is scored 1-4. The total score is achieved by summarizing the score on each question, resulting in a score between 6 and 24. Higher value indicates better health status.
Absolute Claudication Distance (ACD) | Change from Baseline to Up to 6 Months
  ACD is defined as the walking distance after which a patient had to stop walking to relieve claudication pain. Distance is measured in meters
Functional Claudication Distance (FCD) | Change from Baseline to Up to 6 Months
  FCD is defined as the distance a patient would prefer to stop because of claudication pain. Distance is measured in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Gupta, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States